CLINICAL TRIAL: NCT00169195
Title: Gemcitabine-oxaliplatin Plus Rituximab (R-GEMOX) in Refractory/Relapsed Patients With CD 20 Positive Diffuse Large B-cell Lymphoma, Non Eligible for High-dose Chemotherapy Followed by Autotransplantation
Brief Title: Rituximab, Gemcitabine and Oxaliplatin (R-GEMOX) for Refractory/Relapsed B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Hoffmann-La Roche (Industry); Sanofi-Synthelabo (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-GEMOX
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Diffuse Large Cell Lymphoma
Keywords: B-cell lymphoma; Salvage Therapy; rituximab; oxaliplatine; gemcitabine
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — gemcitabine-oxaliplatin regimen; Rituximab

ARMS (1):
- R-GEMOX (Experimental): Gemcitabine-Oxaliplatin plus Rituximab (R-GEMOX)
  Interventions: Drug: Gemcitabine-Oxaliplatin plus Rituximab (R-GEMOX)

INTERVENTIONS:
Drug: Gemcitabine-Oxaliplatin plus Rituximab (R-GEMOX)

SUMMARY:
The Purpose of this study is to evaluate the efficacy and the safety of R-GEMOX in refractory/relapsed patients with CD20-positive large B-cell lymphoma who are not eligible for autologous transplantation.

DETAILED DESCRIPTION:
This is a multicentric, open-label, non-randomized clinical study, evaluating the efficacy and the safety of R-GEMOX in refractory/relapsed patients aged from 18 to 75 years with CD20-positive large B-cell lymphoma non eligible for autologous transplantation.

It is anticipated that 50 subjects will be enrolled over 4 years (from April 2003/January 2007), but inclusion could stop earlier according to the analysis performed every 5 patients (based on triangular test).

The duration of the treatment period is approximately 16 weeks and patients are followed until death.

The total duration of the study is expected to be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with histologically or cytologically proven, CD 20+, diffuse large B-cell lymphoma,
* Relapse after first or second CR, PR or less than PR to first-line treatment for the rituximab-naïve patients, OR relapse after first or second CR with a minimum delay of 12 months between the last rituximab infusion and the inclusion for the rituximab-experienced patients
* Aged 18 - 75 years
* Not eligible for autologous transplantation
* Previously treated with chemotherapy containing anthracycline, with or without rituximab
* ECOG performance status 0 to 2
* With a minimum life expectancy of 3 months
* Having signed informed consent form prior to enrollment

Exclusion Criteria:

* Burkitt's, mantle cell, T-cell lymphomas
* CD 20-negative lymphoma
* HIV or HBV related disease
* Central nervous system or meningeal involvement by the lymphoma
* Not previously treated with anthracycline-containing regimens
* Contraindication to any drug contained in the R-GEMOX chemotherapy regimen
* Any serious active disease or co-morbid medical condition (according to the investigator's decision),
* Poor renal function (creatinine level > 150micromol/l), poor hepatic function (total bilirubin level > 30mmol/l, transaminases > 2.5 maximum normal level) unless these abnormalities are related to the lymphoma
* Poor bone marrow reserve as defined by neutrophils < 1.5 G/l or platelets < 100 G/l, unless related to bone marrow infiltration
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study
* Any radiotherapy during the four weeks before inclusion
* Pregnant or lactating woman
* Adult patient unable to give informed consent because of intellectual impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) (complete response, [CR]; unconfirmed complete response, [CRu] and partial response, [PR]) | 8 weeks
  4 cycles of R-GEMOX

SECONDARY OUTCOMES:
Overall response rate (ORR) (complete response, [CR]; unconfirmed complete response, [CRu] and partial response, [PR]) | 16 weeks
  completion of the treatment
Event free survival (EFS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Haioun, MD, Study Chair — Hôpital Henri Mondor, Créteil, France; Corinne Haioun, MD, Principal Investigator — Hôpital henri Mondor, Créteil, France
Locations (8):
- France (8):
  - Hôpital Henri Mondor, Créteil
  - Service d'Hématologie Clinique - CHU Le Bocage, Dijon
  - Service des Maladies du Sang - CHRU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Saint Louis, Paris
  - Service D'Hématologie Adulte - Hôpital Necker, Paris
  - Centre Henri Becquerel, Rouen
  - CHRU de Nancy Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Chau I, Webb A, Cunningham D, Hill M, Rao S, Ageli S, Norman A, Gill K, Howard A, Catovsky D. An oxaliplatin-based chemotherapy in patients with relapsed or refractory intermediate and high-grade non-Hodgkin's lymphoma. Br J Haematol. 2001 Dec;115(4):786-92. doi: 10.1046/j.1365-2141.2001.03181.x. PMID 11843810
- [Background] Machover D, Delmas-Marsalet B, Misra SC, Gumus Y, Goldschmidt E, Schilf A, Frenoy N, Emile JF, Debuire B, Guettier C, Farrokhi P, Boulefdaoui B, Norol F, Parquet N, Ulusakarya A, Jasmin C. Dexamethasone, high-dose cytarabine, and oxaliplatin (DHAOx) as salvage treatment for patients with initially refractory or relapsed non-Hodgkin's lymphoma. Ann Oncol. 2001 Oct;12(10):1439-43. doi: 10.1023/a:1012501305214. PMID 11762817
- [Background] Faivre S, Raymond E, Woynarowski JM, Cvitkovic E. Supraadditive effect of 2',2'-difluorodeoxycytidine (gemcitabine) in combination with oxaliplatin in human cancer cell lines. Cancer Chemother Pharmacol. 1999;44(2):117-23. doi: 10.1007/s002800050955. PMID 10412945
- [Background] Savage DG, Rule SA, Tighe M, Garrett TJ, Oster MW, Lee RT, Ruiz J, Heitjan D, Keohan ML, Flamm M, Johnson SA. Gemcitabine for relapsed or resistant lymphoma. Ann Oncol. 2000 May;11(5):595-7. doi: 10.1023/a:1008307528519. PMID 10907954
- [Derived] Mounier N, El Gnaoui T, Tilly H, Canioni D, Sebban C, Casasnovas RO, Delarue R, Sonet A, Beaussart P, Petrella T, Castaigne S, Bologna S, Salles G, Rahmouni A, Gaulard P, Haioun C. Rituximab plus gemcitabine and oxaliplatin in patients with refractory/relapsed diffuse large B-cell lymphoma who are not candidates for high-dose therapy. A phase II Lymphoma Study Association trial. Haematologica. 2013 Nov;98(11):1726-31. doi: 10.3324/haematol.2013.090597. Epub 2013 Jun 10. PMID 23753028
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org